CLINICAL TRIAL: NCT02661997
Title: Novel Interventions for Gulf War Veterans' Illnesses
Brief Title: Novel Interventions for GWVI
Acronym: NIGWVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Boston University (Other); Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLD-004-15S
Record Dates: First submitted 2016-01-14; First posted 2016-01-25 (Estimated); Results first posted 2024-11-07 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Gulf War Veteran's Illness
Keywords: Tai Chi; Wellness; Mind-body; Gulf War Illness; Gulf War Veteran's Illness; GWVI

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi Intervention (Experimental): All components of the program derive from the classical Yang Tai Chi 108 postures, which has been shown to be a moderate intensity exercise. Each Tai Chi session will last 60 minutes, twice a week for 12 weeks. In the first session, the Tai Chi instructors will explain exercise theory and procedures of Tai Chi. In subsequent sessions, subjects will practice Tai Chi under the instruction of one of the Tai Chi instructors. Every session will include the following components: (1) warm up and a review of Tai Chi principles; (2) meditation with Tai Chi movement; (3) breathing techniques; and (4) relaxation. The investigators will instruct patients to practice at least 30 minutes a day at home throughout the intervention period and will provide them with training materials for home practice.
  Interventions: Behavioral: Tai Chi Intervention
- Wellness Intervention (Active Comparator): The investigators will utilize a wellness education program for the control group because this approach has been successfully used in other Tai Chi studies from the investigators' team. Participants in the Wellness condition will also attend two 60-minute sessions per week for 12 weeks. The Wellness condition will correspond to the VA Whole Health Program to emphasize wellness across various domains (e.g., physical, emotional, and spiritual lives.) Each session will include a video clip as well as a brief mindfulness exercise that corresponds with the material being presented. The project coordinator for this study will provide the didactic lessons.
  Interventions: Behavioral: Wellness Intervention

INTERVENTIONS:
Behavioral: Tai Chi Intervention — All components of the program derive from the classical Yang Tai Chi 108 postures, which has been shown to be a moderate intensity exercise. Each Tai Chi session will last 60 minutes, twice a week for 12 weeks. In the first session, the Tai Chi instructors will explain exercise theory and procedures of Tai Chi. In subsequent sessions, subjects will practice Tai Chi under the instruction of one of the Tai Chi instructors. Every session will include the following components: (1) warm up and a review of Tai Chi principles; (2) meditation with Tai Chi movement; (3) breathing techniques; and (4) relaxation. The investigators will instruct patients to practice at least 30 minutes a day at home throughout the intervention period and will provide them with training materials for home practice.
  Arms: Tai Chi Intervention
Behavioral: Wellness Intervention — The investigators will utilize a wellness education program for the control group because this approach has been successfully used in other Tai Chi studies from the investigators' team. Participants in the Wellness condition will also attend two 60-minute sessions per week for 12 weeks. The Wellness condition will correspond to the VA Whole Health Program to emphasize wellness across various domains (e.g., physical, emotional, and spiritual lives.) Each session will include a video clip as well as a brief mindfulness exercise that corresponds with the material being presented. The project coordinator for this study will provide the didactic lessons.
  Arms: Wellness Intervention

SUMMARY:
The primary aim of this study was to examine the beneficial effects of two novel treatments for Gulf War Veteran's Illness (Tai Chi and Wellness intervention) and to establish the efficacy of these mind-body approaches to symptom reduction.

In March 2020 after 53 Veterans were randomized, this trial was halted due to the onset of COVID-19. In late 2020, we shifted from conducting an in-person study to a fully remote study with interventions delivered via synchronous video teleconferencing. We then randomized an additional 61 Veterans for a study grand total of 114 Veterans.

DETAILED DESCRIPTION:
Objectives: Over 40,000 Veterans who served in the 1991 Gulf War (GW) have a persistent form of chronic multisymptom illness that defines Gulf War Veterans Illness (GWVI). With no existing proven treatments to provide relief to these sufferers, it is critical to find efficacious and acceptable treatments for GWVI.

The long-term goal was to develop a safe, readily available, mind-body treatment to reduce pain and other chronic symptoms and enhance wellness in Veterans with GWVI. Tai Chi is a traditional Chinese mind-body therapy that has been practiced for centuries. In the last decade, the investigators have demonstrated that Tai Chi can improve both physical health and psychological wellbeing in patients with a variety of chronic conditions.

This randomized trial aimed to establish the effectiveness of a Tai Chi mind-body treatment in Veterans with GWVI. One hundred and fourteen participants meeting criteria for GWVI were randomly assigned to either a Tai Chi exercise or a wellness education group for 12 weeks with a post treatment assessment, and follow-up assessments. The investigators addressed the following Specific Aims:

Specific Aim 1: Evaluate whether the Tai Chi intervention will reduce symptoms of pain in Veterans with GWVI more than the Wellness intervention. The investigators hypothesized that participants randomized to the Tai Chi intervention will show a greater reduction in pain symptoms than those in the Wellness intervention and will maintain changes over a 9-month follow-up period.

Specific Aim 2: Evaluate whether the Tai Chi intervention improves fatigue, cognition, quality of life, and physical functioning in GW Veterans with GWVI, as compared to the Wellness intervention. The investigators hypothesized that participants randomized to the Tai Chi intervention will evidence more improvement in fatigue, cognitive functioning, quality of life, and physical functioning than those randomized to the Wellness intervention and will maintain changes over a 9-month follow-up period.

Research Design: One hundred and fourteen GW Veterans meeting criteria for GWVI were randomly assigned to either the Tai Chi Condition (n=58) or the Wellness Condition (n=56).

Methodology: Participants received 12 weeks of the randomly-assigned intervention twice each week. Assessments were conducted at baseline, 12 weeks (post-intervention), 24 weeks (3 months post-intervention) and 48 weeks (9 months post-intervention). Assessments included instruments to measure self-reported pain, fatigue, cognition, quality of life, and physical functioning.

ELIGIBILITY:
Inclusion Criteria:

* Served in the 1991 Gulf War.
* Meets criteria for chronic multisymptom illness (CMI) based on CDC criteria32 characterized by one or more symptoms of at least 6 months duration from at least two of three symptom categories: 1) musculoskeletal pain (muscle pain, joint pain, or stiffness); 2) fatigue; and 3) mood-cognition.
* One symptom of CMI must be musculoskeletal or joint pain or stiffness of at least 6 months duration (in addition to fatigue or cognitive complaints of the CDC criteria32).
* Not planning to relocate in next 3 months
* English-Speaking: English is the only language to be used during the exercise training program. Our self-reported outcome measures are obtained from validated English-version questionnaires. In addition, using other languages would likely require separate classes, recruitment and instructors which are beyond our current study scope.
* Has access to a home computer or device that will allow telehealth delivery of the intervention.

Exclusion Criteria:

* Lacks the capacity to provide consent
* Major medical, psychiatric, or neurological disorder or has a moderate or severe traumatic brain injury, which could interfere with their ability to safely engage in Tai Chi exercises.
* Change in psychotropic or pain medication during the past month

  * This will minimize amount of symptom change due to medication alterations
  * Once enrolled, medication changes are nonetheless expected and will be monitored
* Regular current Tai Chi, mindfulness, or yoga practice, defined as at least three hours per week for more than three months.

  * Veterans with prior experience who do not currently engage in regular practice at this level will be eligible
* Reports difficulty standing on feet for the majority of a Tai Chi class (approximately 60 minutes).
* Participants who are disruptive or disrespectful or engage in behavior that threatens staff and/or participant safety may be terminated from the study.
* Participants who are currently involved in another treatment study that might confound our findings (e.g., treatments for GWI, pain).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L. Niles, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA; DeAnna L Mori, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niles BL, Grossman S, McQuade M, Grossman D, Kaiser AP, Muccio B, Warner B, Wang C, Mori DL. Study protocol for a revised randomized trial: Remotely delivered Tai Chi and wellness for Gulf War illness. Contemp Clin Trials. 2023 Feb;125:107045. doi: 10.1016/j.cct.2022.107045. Epub 2022 Dec 6. PMID 36494045
- See also: IRB approved webpage - Novel Interventions for Gulf War Illness study — https://www.research.va.gov/for_veterans/gw-holistic.cfm

RESULTS

PARTICIPANT FLOW:
Period: Baseline Assessment
Arm/Group | Tai Chi Intervention | Wellness Intervention
Started | 58 | 56
Completed | 58 | 56
Not Completed | 0 | 0
Period: Post-Treatment Assessment
Arm/Group | Tai Chi Intervention | Wellness Intervention
Started | 58 (We attempted to contact all 114 participants at each assessment point, which is why we indicated 114 started at each timepoint. We think this best represents our methodology. For example, a participant may have completed the baseline, but not the post-treatment assessment, and then completed the 3 and 9-month assessments.) | 56 (We attempted to contact all 114 participants at each assessment point, which is why we indicated 114 started at each timepoint. We think this best represents our methodology. For example, a participant may have completed the baseline, but not the post-treatment assessment, and then completed the 3 and 9-month assessments.)
Completed | 48 | 50
Not Completed | 10 | 6
Period: 3-month Follow-up Assessment
Arm/Group | Tai Chi Intervention | Wellness Intervention
Started | 58 (We attempted to contact all 114 participants at each assessment point, which is why we indicated 114 started at each timepoint. We think this best represents our methodology. For example, a participant may have completed the baseline, but not the post-treatment assessment, and then completed the 3 and 9-month assessments.) | 56 (We attempted to contact all 114 participants at each assessment point, which is why we indicated 114 started at each timepoint. We think this best represents our methodology. For example, a participant may have completed the baseline, but not the post-treatment assessment, and then completed the 3 and 9-month assessments.)
Completed | 52 | 50
Not Completed | 6 | 6
Period: 9-month Follow-up Assessment
Arm/Group | Tai Chi Intervention | Wellness Intervention
Started | 58 (We attempted to contact all 114 participants at each assessment point, which is why we indicated 114 started at each timepoint. We think this best represents our methodology. For example, a participant may have completed the baseline, but not the post-treatment assessment, and then completed the 3 and 9-month assessments.) | 56 (We attempted to contact all 114 participants at each assessment point, which is why we indicated 114 started at each timepoint. We think this best represents our methodology. For example, a participant may have completed the baseline, but not the post-treatment assessment, and then completed the 3 and 9-month assessments.)
Completed | 45 | 46
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi Intervention | Wellness Intervention | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.09 (8.40) | 56.50 (7.41) | 56.80 (7.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 48 | 46 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 18 | 24
  White | 45 | 31 | 76
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Pain Inventory - Short Form (BPI) - Pain Interference
Description: The Brief Pain Inventory (BPI) is a self-report measure that examines pain severity and interference with functioning in various life domains, including general activity, mood, walking activity, work, relationships, sleep, and enjoyment of life. In addition, the BPI asks questions about pain relief, pain quality, and patient perception of the cause of pain. It has been used and validated in a wide range of clinical conditions and is a gold standard measure for the assessment of pain and its impact. Test-retest reliability has been studied in a variety of pain populations and ranges from .83 to .98. Results of the Pain Interference subscale are reported below. Each item of the 7-item subscale is rated from 0 to 10 with higher scores reflecting a worse outcome. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 0 and a maximum score of 10.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
score on a scale
  Baseline Measure | 4.47 (2.69) | 4.77 (2.85)
  Post-Treatment (12 weeks) | 3.59 (2.92) | 3.66 (2.62)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.58, ANOVA — Between group differences

2. Primary Outcome: Change in Brief Pain Inventory - Short Form (BPI) - Pain Severity
Description: The Brief Pain Inventory (BPI) is a self-report measure that examines pain severity and interference with functioning in various life domains, including general activity, mood, walking activity, work, relationships, sleep, and enjoyment of life. In addition, the BPI asks questions about pain relief, pain quality, and patient perception of the cause of pain. It has been used and validated in a wide range of clinical conditions and is a gold standard measure for the assessment of pain and its impact. Test-retest reliability has been studied in a variety of pain populations and ranges from .83 to .98. Results of the Pain Severity subscale are reported below. Each item of the 4-item subscale is rated from 0 to 10 with higher scores reflecting a worse outcome. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 0 and a maximum score of 10.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
score on a scale
  Baseline Measure | 4.28 (1.94) | 4.75 (2.38)
  Post-Treatment (12 weeks) | 4.02 (2.51) | 4.43 (2.46)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.88, ANOVA

3. Secondary Outcome: Change in Multi-dimensional Fatigue Inventory (MFI-20)
Description: The Multidimensional Fatigue Inventory (MFI-20) is a widely-used self-report measure that quantifies symptoms of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Internal consistency and test-retest reliability are strong for all subscales. Responses are made on a 5-point scale from 1-5, with higher scores reflecting greater fatigue. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 1 and a maximum score of 5. Results from the General Fatigue Subscale are provided below.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
score on a scale
  Baseline Measure | 3.62 (1.04) | 3.72 (0.91)
  Post-Treatment (12 weeks) | 3.55 (1.06) | 3.42 (0.93)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.17, ANOVA

4. Secondary Outcome: PROMIS Global Health Scale - Physical Health Subscale
Description: The PROMIS initiative developed new ways to measure patient-reported outcomes such as pain, fatigue, physical functioning, emotional distress, and social role participation that have a major impact on quality-of-life across a variety of chronic diseases. The PROMIS Global Health Scale asks participants to rate their health in terms of physical health, mental health, and satisfaction with social activities, and two scores are produced: Physical Health and Mental Health. Results from the Physical Health Subscale are presented below. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 1 and a maximum score of 5. Higher scores reflect a better outcome.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 92 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 44 | 48
score on a scale
  Baseline Measure | 2.88 (0.70) | 2.93 (0.74)
  Post-Treatment (12 weeks) | 3.00 (0.80) | 3.02 (0.74)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; This is an analysis of pre to post-treatment changes on the Physical Health subscale of the PROMIS Global Health Scale; Test type: Superiority; p = 0.88, ANOVA

5. Secondary Outcome: 50 Foot Walk Test
Description: The Walk 50FT is a widely used timed measure of fast walking speed. It involves a participant walking 50 feet without any use of an aid while study staff monitor and record their time in seconds using a stopwatch. Participants are instructed to walk "as fast as possible." Two trials of the Walk 50FT were conducted and an average score of these two trials was produced. A lower Walk 50FT score is indicative of higher (i.e., faster) walking speed. The Walk 50FT is empirically supported, possesses strong validity and reliability, and demonstrates sensitivity to change over time among individuals with chronic disorders and is a promising measure of physical functioning in patients with a pain-related condition.
Time Frame: Change from baseline to post-treatment (12 weeks)
Population: 98 Veterans participated in the post-treatment assessment, however only 42 completed full data on this measure. This measure could not be administered when the study changed to be a fully remote study during the pandemic.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 20 | 22
seconds
  Baseline measure | 10.72 (2.26) | 10.55 (3.96)
  Post-treatment (12-weeks) | 11.27 (4.04) | 9.64 (2.74)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.032, ANOVA — P-value for group by time interaction

6. Secondary Outcome: Change in Trail Making Test (TMT) - Trails A
Description: The Trail Making Test (TMT) is one of the most popular neuropsychological tests and provides information on visual search, scanning, speed of processing, mental flexibility, and executive functioning. It consists of two parts: A and B. Part A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task B requires a similar task, however a participant is asked to draw a line alternating between numbers and letters (e.g., 1, A, 2, B, 3, C, etc). The score on each part represents the amount of time required to complete the task with higher scores reflecting a worse outcome. Results from Trails A are presented below.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 20 | 22
seconds
  Baseline measure | 25.28 (8.67) | 27.96 (9.34)
  Post-treatment (12-weeks) | 24.75 (8.83) | 26.29 (10.63)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.44, ANOVA — P-value for group by time interaction

7. Secondary Outcome: Change in Trail Making Test (TMT) - Trails B
Description: The Trail Making Test (TMT) is one of the most popular neuropsychological tests and provides information on visual search, scanning, speed of processing, mental flexibility, and executive functioning. It consists of two parts: A and B. Trails A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Trails B requires a similar task, however a participant is asked to draw a line alternating between numbers and letters (e.g., 1, A, 2, B, 3, C, etc). The score on each part represents the amount of time required to complete the task with higher scores reflecting a worse outcome. Results from Trails B is reported below.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 40 completed full data on this measure. This measure could not be administered when the study changed to be a fully remote study during the pandemic.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 19 | 21
seconds
  Baseline measure | 65.91 (30.25) | 63.52 (24.21)
  Post-treatment (12-weeks) | 66.04 (42.60) | 60.52 (24.16)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.73, ANOVA — P-value for group by time interaction

8. Secondary Outcome: Change in Hopkins Verbal Learning Test - Revised (HVLT-R)
Description: The Hopkins Verbal Learning Test- Revised (HVLT-R) is a cognitive test of verbal learning and memory task where participants are instructed to learn a list of 12 nouns over three learning trials. Each time study staff read the list of words, participants are asked to recall as many words from the list as they can remember immediately afterwards. The sum of correctly recalled words over the three trials is a measure of total recall. Scores can range from 0 to 36 with higher scores reflect better a better outcome.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: total words recalled
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 20 | 22
total words recalled
  Baseline measure | 22.25 (4.32) | 21.27 (4.10)
  Post-treatment (12-weeks) | 23.85 (3.91) | 22.59 (4.71)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.36, ANOVA — P-value for group by time interaction

9. Secondary Outcome: PROMIS Global Health Scale - Mental Health Subscale
Description: The PROMIS initiative developed new ways to measure patient-reported outcomes such as pain, fatigue, physical functioning, emotional distress, and social role participation that have a major impact on quality-of-life across a variety of chronic diseases. The PROMIS Global Health Scale asks participants to rate their health in terms of physical health, mental health, and satisfaction with social activities, and two scores are produced: Physical Health and Mental Health. Results from the Mental Health Subscale are presented below. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 1 and a maximum score of 5. Higher scores reflect a better outcome.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 92 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Wellness Intervention: Wellness Intervention: The investigators will utilize a wellness education program for the control group because this approach has been successfully used in other Tai Chi studies from the investigators' team. Participants in the Wellness condition will also attend two 60-minute sessions per week for 12 weeks. The Wellness condition will correspond to the VA Whole Health Program to emphasize wellness across various domains (e.g., physical, emotional, and spiritual lives.) Each session will include a video clip as well as a brief mindfulness exercise that corresponds with the material being presented.
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 44 | 48
units on a scale
  Baseline Measure | 2.44 (0.93) | 2.67 (0.84)
  Post-treatment Measure (12-weeks) | 2.73 (1.11) | 2.83 (0.82)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.24, ANOVA

10. Secondary Outcome: Short Physical Performance Battery (SPPB) - 4-Meter Walk Test
Description: The Short Physical Performance Battery (SPPB) captures domains of strength, endurance, and balance and is highly predictive of disability. The SPPB is based on three timed measures of standing balance, walking (gait) speed, and ability to rise from a chair. The 4-Meter Walk Test is a measure of gate speed where participants are asked to walk 4-meters at a normal walking pace while being timed. Results from the 4-Meter Walk Test are presented below.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 20 | 22
seconds
  Baseline measure | 5.26 (1.14) | 5.54 (0.92)
  Post-treatment (12-weeks) | 5.23 (1.19) | 4.70 (1.02)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.006, ANOVA — P-value for group by time interaction

11. Secondary Outcome: Short Physical Performance Battery (SPPB) - Chair Stand Test (CST)
Description: The Short Physical Performance Battery (SPPB) captures domains of strength, endurance, and balance and is highly predictive of disability. The SPPB consists of three timed measures: standing balance, walking speed, and ability to rise from a chair. The Chair Sit Test (CST) is a timed evaluation of the strength and power of lower-extremities. Participants are instructed to complete five chair stands from a sitting position with their arms folded across their chests. They are instructed to do this as fast as possible, while being timed. Lower scores reflect a better outcome.
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 39 completed full data on this measure. This measure could not be administered when the study changed to be a fully remote study during the pandemic.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 18 | 21
seconds
  Baseline measure | 13.60 (3.13) | 12.49 (3.39)
  Post-treatment (12-weeks) | 13.92 (5.03) | 13.20 (7.94)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.55, ANOVA — P-value for group by time interaction

12. Secondary Outcome: Short Physical Performance Battery (SPPB) - Standing Balance Test (SBT)
Description: The SPPB captures domains of strength, endurance, and balance and is highly predictive of disability. The SPPB consists of three timed measures: standing balance, walking speed, and ability to rise from a chair. The Standing Balance Test measures ability to balance while holding in three different positions for 10 seconds. For each position they are able to hold for 10 seconds, they receive a score of 1. If they are unable to hold the position, they receive a score of 0. To illustrate the minimal variability on this measure, results are provided below for the tandem position (the most difficult position to hold).
Time Frame: Change from baseline to post-treatment at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 41 completed full data on this measure. This measure could not be administered when the study changed to be a fully remote study during the pandemic.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 19 | 22
units on a scale
  Baseline measure | 1.0 (0) | 1.0 (0)
  Post-treatment (12-weeks) | 1.0 (0) | .95 (.21)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.36, ANOVA — P-value for group by time interaction

13. Other Pre Specified Outcome: Health Symptom Checklist (HSC)
Description: The Health Symptom Checklist consists of 34 frequently reported health and mental health symptoms from nine body systems (cardiac, pulmonary, dermatological, gastrointestinal, genitourinary, musculoskeletal, neurological, neuropsychological and psychological). On a 5 point scale from 0 (no) to 4 (very often), respondents indicate if they have experienced each symptom in the last 30 days, and if yes, how often. A response of 2 (about once per week) or greater is considered an endorsement of the symptom. All symptoms endorsed are added together for a total score. Total scores can range from 0 to 34 with higher scores indicating more symptoms.
Time Frame: Change from baseline HSC at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
score on a scale
  Baseline Measure | 18.82 (7.87) | 17.53 (8.35)
  Post-treatment | 18.07 (8.37) | 15.27 (8.38)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.13, ANOVA

14. Other Pre Specified Outcome: The PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5) is a self-report measure consisting of 20 items that parallel the DSM-5 posttraumatic stress disorder criteria. Respondents indicate on a 5-point scale (0-4) how much they have been bothered in the last month by particular symptoms that are related to stressful military experiences. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 0 and a maximum score of 4.The DSM-IV version of the PCL has been shown to have excellent reliability and validity.
Time Frame: Change from baseline PCL-5 at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
units on a scale
  Baseline Measure | 1.85 (1.04) | 1.86 (1.02)
  Post-treatment | 1.72 (1.01) | 1.60 (0.96)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.26, ANOVA

15. Other Pre Specified Outcome: Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. It is comprised of seven questions that are responded to on a scale from 0 to 4.. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 0 and a maximum score of 4, with higher scores reflecting greater insomnia symptom severity.
Time Frame: Change from baseline ISI at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 86 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 43
units on a scale | 2.40 (1.11) | 2.38 (0.90)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.04, ANOVA

16. Other Pre Specified Outcome: Participant Compliance Log - Intervention Sessions Attended
Description: Study staff will monitor number of intervention sessions attended. The maximum total number of sessions is 24 (range 0-24) with higher numbers showing greater number of sessions attended.
Time Frame: 12 weeks
Population: This data was collected on all 114 participants who were validly randomized for this study.
Measure: Mean (Standard Deviation); unit: sessions attended
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 58 | 56
sessions attended | 15.62 (7.33) | 16.95 (7.62)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.35, t-test, 2 sided

17. Other Pre Specified Outcome: Participant Compliance Log - Assessment Sessions Attended
Description: Percentage of participants who completed the post-treatment assessment.
Time Frame: 12 weeks
Population: This data was collected on all 114 participants who were validly randomized for this study.
Measure: Number; unit: percentage of participants
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 58 | 56
percentage of participants | 82.8 | 89.3

18. Other Pre Specified Outcome: Weekly Practice Log Sheet
Description: This measure will monitor compliance with home Tai Chi practice during the intervention. Average Tai Chi practice minutes per week is reported.
Time Frame: 12 weeks
Population: 58 Veterans were randomized to Tai Chi, however only 54 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Tai Chi Intervention
Number analyzed (Participants) | 54
minutes per week | 183.62 (87.70)

19. Other Pre Specified Outcome: Client Satisfaction Questionnaire
Description: The Client Satisfaction Questionnaire (CSQ) is is an 8-item measure that assesses satisfaction with both the interventions. Each item is responded to on a 4-point scale (1-4) and items are summed for a total score that can range from 8-32 with higher scores reflecting greater satisfaction.
Time Frame: Difference between two intervention groups at post-treatment (12 weeks)
Population: 98 Veterans participated in the post-treatment assessment, however only 87 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 42 | 45
units on a scale | 28.81 (3.64) | 27.67 (3.74)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.15, t-test, 2 sided

20. Other Pre Specified Outcome: Depression Anxiety Sensitivity Scale (DASS) - Depression Scale
Description: The Depression Anxiety Sensitivity Scale (DASS) is a 21 item questionnaire that is responded to on a 4-point scale that ranges from 0-3. There are three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. Scores are obtained by summing the items that comprise each of the three scales, with higher scores reflecting greater symptomatology. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 0 and a maximum score of 3.The DASS was constructed not merely as another set of scales to measure conventionally defined emotional states, but to further the process of defining, understanding, and measuring the ubiquitous and clinically significant emotional states usually described as depression, anxiety and stress.
Time Frame: Change from baseline DASS at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 92 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 44 | 48
units on a scale
  Baseline Measure | 1.18 (0.90) | 1.03 (0.87)
  Post-treatment | 0.95 (0.97) | 0.82 (0.74)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.91, ANOVA

21. Other Pre Specified Outcome: Depression Anxiety Sensitivity Scale (DASS) - Anxiety Scale
Description: as for outcome 20
Time Frame: Change from baseline DASS at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 92 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 44 | 48
units on a scale
  Baseline Measure | 0.95 (0.73) | 0.86 (0.66)
  Post-treatment | 0.85 (0.75) | 0.69 (0.62)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.42, ANOVA

22. Other Pre Specified Outcome: Depression Anxiety Sensitivity Scale (DASS) - Stress Scale
Description: as for outcome 20
Time Frame: Change from baseline DASS at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 92 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 44 | 48
units on a scale
  Baseline Measure | 1.21 (0.73) | 1.36 (0.69)
  Post-treatment | 1.14 (0.81) | 1.12 (0.70)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.10, ANOVA

23. Other Pre Specified Outcome: Change in the Pain Catastrophizing Scale (PCS)
Description: The PCS is a 13-item self-report scale that assesses the degree to which people engage in three subtypes of pain catastrophizing: rumination, magnification, and helplessness. Each item is responded to on a 5 point scale (0-4). Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 0 and a maximum score of 4, with higher scores reflecting greater pain catastrophizing. It is one of the most widely used instruments for measuring catastrophic thinking in relation to pain.
Time Frame: Change from baseline PCS at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 89 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 44 | 45
units on a scale
  Baseline Measure | 1.61 (1.10) | 1.49 (1.16)
  Post-treatment | 1.43 (0.99) | 1.31 (1.05)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.99, ANOVA

24. Other Pre Specified Outcome: Change in West Haven-Yale Multidimensional Pain Inventory (WHYMPI) - General Activity Scale
Description: The West Haven-Yale Multidimensional Pain Inventory (WHMPI) is a well-validated measure of the experience of chronic pain and has been shown to be applicable across a variety of clinical pain conditions. The 52-item inventory is divided into three parts: 1) Important dimensions of the chronic pain experience, 2) patient perceptions of how important others respond to their pain, and 3) engagement in everyday activities. Patient's responses to WHYMPI items are made on a 7-point scale (0-6). The focus of the analysis reported before is on the 18 items that constitute Part 3. This General Activity Scale was scored by summing responses and then obtaining an average by dividing by the number of non-missing items. Total average scores range from 0-6 with higher scores reflecting greater engagement in common everyday activities.
Time Frame: Change from baseline WHYMPI at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
units on a scale
  Baseline Measure | 2.84 (1.06) | 2.58 (0.94)
  Post-treatment | 2.76 (1.00) | 2.80 (1.07)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.09, ANOVA

25. Other Pre Specified Outcome: Change in Chronic Pain Self-Efficacy Scale (CPSS)
Description: The Chronic Pain Self-Efficacy Scale (CPSS) is a 22-item questionnaire designed to measure chronic pain patients' perceived self-efficacy to cope with the consequences of chronic pain. Questions are broken down into three categories: self-efficacy for pain management, self-efficacy for physical function, and self-efficacy for coping with symptoms. Each item in the CPSS is presented as a question (e.g., "How certain are you that you can decrease your pain quite a bit?"). Participants rate each belief on a 10-point Likert scale (range 10-100). A total score is calculated by first summing the item responses across all three categories. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 10 and a maximum score of 100, with higher scores reflecting greater perceived self-efficacy.
Time Frame: Change from baseline CPSS at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
units on a scale
  Baseline Measure | 61.09 (18.60) | 57.25 (18.45)
  Post-treatment | 63.02 (18.81) | 61.52 (19.94)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.44, ANOVA

26. Other Pre Specified Outcome: Group Cohesiveness Scale (GSC)
Description: The Group Cohesiveness Scale is a self-report measure that examines group cohesion within a therapeutic environment. Each of the 7 questions are responded to on a 5-point scale (1-5). Scores are obtained by summing the items with higher scores reflecting greater group cohesiveness.
Time Frame: Post-treatment measure taken at 12 weeks
Population: 72 Veterans participated in this week 12 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 33 | 39
units on a scale | 28.12 (6.47) | 30.49 (4.67)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.09, t-test, 2 sided — An adjusted p value was used based on Levene's test

27. Other Pre Specified Outcome: PROMIS Self-Efficacy for Managing Symptoms
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Symptoms is an 8-item self-report measure that examines elements of self-care. Each item is responded to on a 5 point scale ranging from 1-5. Raw scores are calculated by summing responses to all the items (score range 8-40), and then converted to a T-score using a conversion table located in the administration guide provided for the PROMIS instruments. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. Higher scores reflect greater confidence in one's ability to manage one's symptoms
Time Frame: Change from baseline PROMIS Self-Efficacy at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 92 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 44 | 48
units on a scale
  Baseline Measure | 45.75 (9.66) | 45.71 (8.08)
  Post-treatment | 46.51 (9.76) | 46.00 (7.70)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.75, ANOVA

28. Other Pre Specified Outcome: Mindfulness Attention Awareness Scale (MAAS)
Description: The Mindfulness Attention Awareness Scale (MAAS) is a 15-item self-report measure that assesses participants' openness towards, awareness of, and attention to the present. This scale can reveal information about one's self-regulation and well-being. Each item is responded to on a 6-point scale from 1 (almost always) to 6 (almost never) with higher scores reflecting greater mindfulness awareness. Sum scores are changed to mean scores so they are in the same metric as the individual items constituting the scale with a minimum score of 1 and a maximum score of 6.
Time Frame: Change from baseline MAAS at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 91 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 43 | 48
units on a scale
  Baseline Measure | 3.85 (1.16) | 3.91 (1.05)
  Post-treatment | 3.99 (1.24) | 4.18 (1.12)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.44, ANOVA

29. Other Pre Specified Outcome: Body Mass Index (BMI)
Description: Study staff recorded participants' height in inches and weight in pounds. Weight and height measurements were used to calculate Body Mass Index using the formula: [weight (lb) / height (in)^2] x 703. This data is only available for the participants who participated in-person.
Time Frame: Change from baseline measurements at 12 weeks
Population: 42 Veterans participated in the in-person post-treatment assessment and all 42 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 20 | 22
kg/m^2
  Baseline Measure | 31.23 (6.03) | 31.43 (4.90)
  Post-treatment | 31.43 (5.95) | 31.87 (4.18)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.67, ANOVA

30. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Systolic pressures were measured in mmHg using a blood pressure cuff and sphygmomanometer. Two blood pressure readings were taken at each assessment point, and the average was used. This data is only available for the participants who were in-person.
Time Frame: Change from baseline measurements at 12 weeks
Population: 42 Veterans participated in the in-person post-treatment assessment and data for all 42 is available on this measure.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 20 | 22
millimeters of mercury
  Baseline Measure | 127.07 (16.05) | 126.64 (11.41)
  Post-treatment | 125.49 (15.18) | 128.92 (13.57)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.43, ANOVA

31. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: Diastolic pressures were measured in mmHg using a blood pressure cuff and sphygmomanometer. Two blood pressure readings were taken at each assessment point, and the average was used. This data is only available for the participants who were in-person.
Time Frame: Change from baseline measurements at 12-weeks
Population: 42 Veterans participated in this in-person post-treatment assessment and data is available for all 42.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 22 | 20
millimeters of mercury
  Baseline Measure | 84.70 (10.79) | 86.33 (9.66)
  Post-treatment | 82.66 (7.75) | 85.23 (11.81)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.80, ANOVA

32. Other Pre Specified Outcome: Physical Activity Recall (PAR) - General Physical Activity
Description: The Physical Activity Recall (PAR) is a measure that was administered by study staff in an interview format. The PAR asks participants' to report time they spent engaged in general physical activity, strength building activities, and activities that involve flexibility over the past week. For the measure of general physical activity, all activity that is of at least moderate intensity is counted and is reported as hours of activity in the past week.
Time Frame: Change from baseline PAR at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 95 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 47 | 48
hours per week
  Baseline Measure | 9.05 (10.34) | 10.55 (9.82)
  Post-treatment | 9.66 (10.95) | 9.11 (9.14)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.31, ANOVA

33. Other Pre Specified Outcome: Physical Activity Recall (PAR) - Strength Activity
Description: The Physical Activity Recall (PAR) is a measure that was administered by study staff in an interview format. The PAR asks participants' to report time they spent engaged in general physical activity, strength building activities, and activities that involve flexibility over the past week. For the measure of strength activity, time spent engaged in strength building activity over the past seven days is totaled and is reported as hours of strength activity in the past week.
Time Frame: Change from baseline PAR Strength time at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 95 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: hours of activity per week
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 47 | 48
hours of activity per week
  Baseline Measure | 0.40 (0.89) | 1.04 (3.95)
  Post-treatment | 0.55 (1.13) | 0.32 (0.89)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.16, ANOVA

34. Other Pre Specified Outcome: Physical Activity Recall (PAR) - Flexibility Activity
Description: The Physical Activity Recall (PAR) is a measure that was administered by study staff in an interview format. The PAR asks participants' to report time they spent engaged in general physical activity, strength building activities, and activities that involve flexibility over the past week. For the measure of flexibility activity, time spent engaged in activity that involve flexibility over the past seven days is totaled and is reported as hours of flexibility activity in the past week.
Time Frame: Change from baseline PAR Flexibility time at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 95 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: Hours of activity per week
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 47 | 48
Hours of activity per week
  Baseline Measure | 0.52 (0.81) | 0.57 (0.94)
  Post-treatment | 1.75 (1.86) | 0.46 (0.77)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p < 0.001, ANOVA

35. Other Pre Specified Outcome: The Epidemic - Pandemic Impacts Inventory (EPII) - Negative Impacts
Description: The Epidemic - Pandemic Impacts Inventory (EPII) is a 92-item questionnaire. This recently-developed measure was designed to learn about and describe the impact of the coronavirus disease pandemic on various domains of personal and family life, including employment, education, home life, social life, economic, physical health, infection experiences, and positive changes. This instrument was only administered to the remote participants, after the pandemic started. Participants were asked to respond to each item with one of the following four responses: 1) "Yes, me", 2) "Yes, person in home", 3) "no", and 4) "not applicable". Any "yes" response was coded as 1 and a "no" or "not applicable" response was coded as 0. Two scales were created (Positive Impacts and Negative Impacts) by summing the items for each scale. Negative Impacts are reported here (possible response range of 0-73), with higher scores indicating greater negative impact of the pandemic.
Time Frame: Change from baseline EPII at 12 weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 50 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 24 | 26
units on a scale
  Baseline Measure | 17.25 (10.66) | 18.58 (8.83)
  Post-treatment | 16.95 (10.61) | 17.29 (8.21)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.56, ANOVA

36. Other Pre Specified Outcome: The Epidemic - Pandemic Impacts Inventory (EPII) - Positive Impacts
Description: The Epidemic - Pandemic Impacts Inventory (EPII) is a 92-item questionnaire. This recently-developed measure was designed to learn about and describe the impact of the coronavirus disease pandemic on various domains of personal and family life, including employment, education, home life, social life, economic, physical health, infection experiences, and positive changes. This instrument was only administered to the remote participants, after the pandemic started. Participants were asked to respond to each item with one of the following four responses: 1) "Yes, me", 2) "Yes, person in home", 3) "no", and 4) "not applicable". Any "yes" response was coded as 1 and a "no" or "not applicable" response was coded as 0. Two scales were created (Positive Impacts and Negative Impacts) by summing the items for each scale. Positive Impacts are reported here (possible response range of 0-18), with higher scores indicating greater positive impact of the pandemic.
Time Frame: Change from baseline EPII at 12 weeks Change from baseline EPII at 12-weeks
Population: 98 Veterans participated in the post-treatment assessment, however only 50 completed full data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi Intervention | Wellness Intervention
Number analyzed (Participants) | 24 | 26
units on a scale
  Baseline Measure | 5.05 (3.53) | 7.38 (4.60)
  Post-treatment | 6.04 (5.01) | 8.83 (4.87)
Statistical Analysis 1: Comparison: Tai Chi Intervention vs Wellness Intervention; Test type: Superiority; p = 0.64, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tai Chi Intervention | Wellness Intervention
All-Cause Mortality (participants affected / at risk) | 1/58 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/58 | 2/56
Other Adverse Events (participants affected / at risk) | 3/58 | 2/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tai Chi Intervention (N=58) | Wellness Intervention (N=56)
Detox from opiates (Psychiatric disorders) | 0 (0) | 1 (1) — Participant sought voluntary hospitalization for detox from opiates
Hospitalization for cardiac symptoms (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tai Chi Intervention (N=58) | Wellness Intervention (N=56)
Blood pressure elevated (Vascular disorders) | 0 (0) | 1 (1)
Cyst on back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Feeling unwell and exhausted (General disorders) | 1 (1) | 0 (0)
Blood sugar elevated (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT02661997/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02661997/ICF_001.pdf